CLINICAL TRIAL: NCT00629096
Title: Effects of Intracoronary Infusion of Bone Marrow-derived Progenitor Cells on Myocardial Regeneration in Patients With Non-ischemic Dilated Cardiomyopathy.
Brief Title: Intracoronary Infusion of Autologous Bone Marrow Cells for Treatment of Idiopathic Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCMR0007/2006; EudraCT 2007-003088-36
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2013-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated Cardiomyopathy; Marrow stem cells; Myocardial regeneration; Mesenchymal stem cells; Marrow-derived endothelial progenitor cells
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All included patients are assigned to arm 1, in which they are treated by the intervention
  Interventions: Procedure: Intracoronary infusion of autologous bone marrow cells

INTERVENTIONS:
Procedure: Intracoronary infusion of autologous bone marrow cells — Autologous mononuclear bone marrow cells will be administered by intracoronary infusion via a percutaneous catheter

SUMMARY:
The main aim of the study is to determine whether intracoronary infusion of autologous bone marrow mononuclear cells can improve the ventricular function of patients with idiopathic dilated cardiomyopathy.Secondary end-points will be:

1. To evaluate possible changes in patient functional capacity and
2. to identify the biological characteristics of the bone marrow graft that might influence on functional recovery.

DETAILED DESCRIPTION:
Clinical studies have shown that bone marrow cells can regenerate damaged myocardium after ischemic cardiopathy; however scarce information is available from patients with non-ischemic dilated cardiomyopathy. The aim of the present work is to investigate the role of intracoronary infusion of autologous marrow-derived stem cells in a phase II study in 30 patients with dilated cardiomyopathy.Before the intracoronary transplant of marrow cells as well as six and twelve months thereafter, we will compare the ventricular function measured as left-ventricular ejection fraction by angiography, magnetic resonance imaging, echocardiography and treadmill direct oxygen consumption test. Functional capacity will be monitored throughout the study. In every condition of the study we will perform at least one 30º right anterior oblique left ventricle (LV)angiogram. During each ventriculogram, attempts will be made to obtain a sinus and a post-extrasystolic beat for analysis, in order to study contractile reserve behaviours. Post-extrasystolic beats will be obtained by inducing premature beats with the catheter, once a well opacified cardiac cycle with a normal sinus beat had been filmed. In all instances, the r-r' interval of the induced premature beat and the post-extrasystolic pause will be recorded and measured.

Measurements and calculations will be made off line in our own core lab, where end-diastolic and end-systolic silhouettes were drawn using the CASS system by 2 expert angiographers who were unaware of the patient group or study conditions. LV-volumes and ejection fraction (EF) were derived and regional wall motion was analyzed. The method by Sheehan (1) was used for the asynergy study, dividing the superimposed silhouettes in 100 radii of wall shortening, from end-diastole to end-systole. The abnormal contracting segment (ACS) was defined as the percentage of radii showing akinesia or dyskinesia. The areas of the ventrivular walls having asynergy will be regionally evaluated. The serial evolution of the contractile reserve will be evaluated by the post-extrasystolic potentiation.

Coronary Flow Reserve (CFR) in all 3 coronary arteries will also be evaluated during every hemodynamic study (before treatment and 6 months after treatment). The FloMap® system (Cardiometrics; Mountain View; California) will be used. A 0.014" intracoronary Doppler guide wire will be positioned proximally in every coronary and flow velocities will be recorded continuously. Average peak velocity will be obtained at baseline and after an intracoronary bolus of Adenosine. CFR will be calculated as the ratio between maximal flow velocity during the peak effect of the adenosine injection and basal flow velocity.

Magnetic Resonance Image (MRI) studies will be performed in 3 conditions (baseline, 3-month and 1-year after treatment). Functional parameters will be obtained in each condition, including LV-volumes, LV-mass and ejection fraction

On the morning of cardiac catheterization, up to a volume of 100-150 ml of marrow will be obtained under local anesthesia by aspiration from the iliac crest. Mononuclear Bone Marrow Cells (MNBMCs) will be isolated by density gradient centrifugation over Ficoll-Hypaque technique in a sterile, semiautomated device COBE® 2991. After three washes, MNBMCs will be filtered and resuspended in 10 ml of 0.9% sodium chloride supplemented with preservative-free 0.1% heparin. Aliquots will be obtained for cell count as well as for cytofluorometric and functional analyses of the cell content.

Cells will be directly transferred to all 3 coronary arteries (50% to left anterior descending artery, 25% to the circumflex and 25% to the right coronary artery) by the use of a coaxial balloon catheter, which will be placed proximally at each artery. Balloon size will be selected according to vessel size, in order to achieve complete occlusion of the vessel and to stop flow during cell injection. So, backflow of cells is prevented and distal stagnant flow will facilitate cell exposure. The cell suspension will be injected through the distal tip of the balloon over 2 to 4 minutes.

In addition,we will try to compare all possible changes in functional parameters with biological variables obtained from the marrow graft, such as:

1. Number of cells positive for cluster of differentiation antigen (CD) CD146,CD31, CD133,CD90,CD38, CD117, CD73, CD105, CD45, Vascular endothelial growth factor receptor 2,CXC-chemokine receptor 4 and HLA-DR.
2. Functional characterization of endothelial progenitor cells and mesenchymal stem cells present in the graft by in vitro selective cultures.
3. Analysis of the in vitro chemotactic ability of the infused cells.
4. Determination of lineage-specific cardiac markers GATA-4 and Nk2.5/Csx in the infused marrow-derived cells. Correlations between these biological parameters and the effects on patient's ventricular function could highlight the role of each of the potential mechanisms implied in cell-mediated myocardial regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with established clinical and angiographic diagnosis of Idiopathic Dilated Cardiomyopathy who accept to participate in the trial.
2. They should have symptoms and/or signs of heart failure, despite optimized medical treatment.
3. Angiographic ejection fraction should be less than 50%.

Exclusion Criteria:

1. Associated coronary artery disease.
2. Any history or suspicion of a toxic, pharmacologic or deposit etiology.
3. Absence of resynchronization therapy.
4. Age longer than 80 years.
5. Associated malignant or pre-malignant systemic disease.
6. Associated hematologic disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Improvement of left ventricular function | 6 and 12 months

SECONDARY OUTCOMES:
Functional status | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Suarez de Lezo, MD, PhD, Study Chair — Department of Cardiology. Reina Sofía University Hospital; I. Concepción Herrera, MD, PhD, Study Director — Department of Hematology.Reina Sofia University Hospital; Manuel Pan, MD, PhD, Principal Investigator — Department of Cardiology. Reina sofia University Hospital; Jose Maria Arizon, MD, Principal Investigator — Department of Cardiology. Reina Sofía university Hospital; Miguel Angel Romero, MD, PhD, Principal Investigator — Department of Cardiology. Reina Sofía University Hospital; Ramon Ribes, MD, PhD, Principal Investigator — Department of Radiology. Reina Sofía University Hospital; Joaquin Sanchez, MD, PhD, Principal Investigator — Department of Hematology. Reina Sofía Unuversity Hospital; Antonio Torrers, MD, PhD, Principal Investigator — Department of Hematology. Reina Sofía University Hospital
Locations (1):
- Reina Sofía University Hospital, Córdoba, Córdoba, Spain